CLINICAL TRIAL: NCT03322228
Title: Music Therapy Intervention to Reduce Caregiver Distress at the End of Life: A Feasibility Study
Brief Title: Music Therapy Intervention to Reduce Caregiver Distress at the End of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Maria I. Lapid, M.D., M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-005811
Record Dates: First submitted 2017-10-13; First posted 2017-10-26 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Quality of Life; Stress; Anxiety; Depression
Keywords: Hospice; Palliative Care; Integrative Medicine; Music Therapy; Inpatient; Caregiver
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: This study plans to enroll 20 subjects. All subjects will receive 1 music therapy intervention lasting approximately 1 hour.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music Therapy (Experimental): 1 music therapy session, lasting approximately 45 min-1 hr
  Interventions: Other: Music Therapy

INTERVENTIONS:
Other: Music Therapy — Music therapy is tailored to subject preference. Examples are active music-making, supportive listening, and includes opportunities for legacy building to decrease caregiver distress and promote self-care.

SUMMARY:
This is a study to assess the feasibility and acceptability of implementing a music therapy intervention for caregivers of hospitalized patients who are referred to inpatient hospice.

DETAILED DESCRIPTION:
Caregivers are at high risk for stress, poor quality of life (QOL), and burnout. As a patient nears death, common themes for caregivers include anxiety and emotional distress from impending death, anticipatory grief, and acceptance of loss, which negatively impact the caregiver QOL. Investigators propose to conduct a pilot project to investigate music therapy impact on caregiver distress for caregivers of imminently dying hospitalized patients referred to hospice. Upon enrollment, caregivers will be provided a music therapy intervention with legacy-building components, and will be asked to complete 3 brief questionnaires on distress and quality of life before and after the music therapy to assess their response to the intervention. The overall aim is to reduce caregiver distress and optimize QOL.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Self-identified caregiver
3. English-speaking

Exclusion Criteria:

1. Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Pearlin role overload measure (ROM) | Baseline to 6 months
  4-item self-administered measure of caregiver stress

SECONDARY OUTCOMES:
Linear Analogue Self-Assessment (LASA) | Baseline to 6 months
  10-item self-report of general measures of quality of life (QOL)
Patient Health Questionnaire for Depression and Anxiety (PHQ-4) | Baseline to 6 months
  4-item self-administered screening tool that combined two validated two-item screeners for depression and anxiety
Music Therapy Program Survey | Up to 72 hours after intervention
  Survey to assess satisfaction regarding the therapy service provided

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lapid, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whitford KJ, Ulrich AM, Larsen BE, Phelps CM, Siska MJ, Bigelow ML, Dockter TJ, Wood C, Walton MP, Stelpflug AJ, Lapid MI. Music Therapy Intervention to Reduce Caregiver Distress at End of Life: A Feasibility Study. J Pain Symptom Manage. 2023 May;65(5):e417-e423. doi: 10.1016/j.jpainsymman.2023.01.009. Epub 2023 Jan 19. PMID 36682675
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials